CLINICAL TRIAL: NCT02809755
Title: Sphenopalatine Ganglion Block to Prevent Shoulder Pain After Laparoscopic Bariatric Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: While 33 people signed consent, no one was enrolled in the study, because none of these patients developed shoulder pain in the recovery room.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-01278
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: Obesity; laparoscopic gastric banding; band revision; laparoscopic gastric banding sleeve gastrectomy
MeSH Terms: conditions — Obesity | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4% lidocaine (Experimental): 10 mL vials filled with 4% lidocaine or normal saline (50 vials of each solution) and pharmacist will code the vials from 1 to 100 using a computer-generated randomization scheme.
  Interventions: Drug: 4% Lidocaine
- Placebo Saline (Placebo Comparator): 10 mL vials filled with 4% lidocaine or normal saline (50 vials of each solution) and pharmacist will code the vials from 1 to 100 using a computer-generated randomization scheme.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: 4% Lidocaine
  Arms: 4% lidocaine
Other: Saline
  Arms: Placebo Saline

SUMMARY:
The purpose of this study is to determine the efficacy of sphenopalatine ganglion (SPG) block to prevent shoulder tip pain following primary laparoscopic gastric banding, band revision, band replacement, primary sleeve gastrectomy or revision of sleeve gastrectomy. Shoulder tip pain (STP) is a common problem after laparoscopic surgery, manifesting in the post-anesthesia care unit and for days or possibly weeks thereafter (Dixon 2005). Systemic analgesics including opioids and non-steroidal anti-inflammatory drugs (NSAIDs) do not reliably relieve STP. This study is designed to determine if the SPG block, a simple and low-risk procedure, effectively treats STP after laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, parallel group prospective, double-blind study. The primary outcome variable will be change in STP from > 4 before to after treatment in the PACU after primary laparoscopic gastric banding, band revision, band replacement, sleeve gastrectomy, or revision of sleeve gastrectomy. Investigators hope to achieve a decline in STP in 2 units after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary laparoscopic gastric banding surgery.
* Laparoscopic band revision surgery
* Laparoscopic band replacement surgery.
* Sleeve gastrectomy.
* Revision of sleeve gastrectomy.
* American Society of Anesthesiologists Class 2 or 3.
* No allergy to study drugs.
* Facility with English language to allow compliance with study protocol.

Exclusion Criteria:

* American Society of Anesthesiologists Class 4 or 5.
* Allergy to lidocaine or to any local anesthetic
* Allergy to oxymetazoline (Afrin)
* Pregnancy
* Bleeding diathesis
* Known nasal pathology including active sinusitis
* Previous nasal surgery
* Preoperative anticoagulant use OTHER THAN aspirin 81 mg and/or heparin 5000 U SQ bid administered for DVT prophylaxis.
* Acute psychiatric disease
* History of chronic right or left shoulder pain
* Current opioid use
* Any patient that the study team feels will be unable to comply with all protocol related procedures
* Concurrent participation in another clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-08; Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Change in STP as assessed by Numeric Rating Scale (NRS-11), from before to after the treatment in the PACU after receiving a 30-minute unilateral SPG block or bilateral SPG block | Baseline, 30 Minutes
  subject will be asked to rate her/his pain from zero to ten with zero being "no pain" to ten being "the worst pain imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Grant, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States